CLINICAL TRIAL: NCT04561609
Title: The Effect of Transcutaneous Application of Gaseous CO2 on Diabetic Chronic Wound Healing
Brief Title: Transcutaneous Application of Gaseous CO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Helena Ban Frangez, assistant professor MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCLjubljana CO2 application
Record Dates: First submitted 2020-09-06; First posted 2020-09-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Wound of the Lower Limb (Leg Ulcer or Foot Ulcer)
Keywords: transcutaneous CO2 application
MeSH Terms: conditions — Leg Ulcer; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: The use of transcutaneous application of gaseous CO2 for treatment of diabetic chronic wound. A Control group receives standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 treated (Active Comparator): Patients receiving treatment with transcutaneous application of gaseous CO2 on lower limbs
  Interventions: Other: Transcutaneous CO2 application
- control (No Intervention): Patients receiving standard of care

INTERVENTIONS:
Other: Transcutaneous CO2 application — Patients lie on examination tables. Lower extremities of the patients are isolated in a therapeutic wrap (single use, low-density, made from biocompatible polyethylene), sealed at the waist. After this, air is first pumped out of the therapeutic wrap, then the wrap was filled with 99.9% CO2 gas. The therapy lasts for 50 minutes.
  Each patient from the study group will receive CO2 therapies - four weeks (meaning 20 CO2 therapies that were performed on workdays only).
  Arms: CO2 treated

SUMMARY:
The research is designed to evaluate influence of transcutaneous application of CO2 (carbon dioxide) on chronic wound healing. Transcutaneous application of CO2 is known to have immediate effect on vasodilatation and elevates oxygen release from Hb via the Bohr effect. After repetition of the therapies neoangiogenesis is induced. Impairment of microcirculation is one of the causes of impared wound healing and improvement in circulation could have positive effect on wound healing, reduction of the wound area and granulation of the wound bed (Falanga score).

DETAILED DESCRIPTION:
Transcutaneous application of gaseous CO2 showed to be a successful adjuvant therapy in treatment of chronic wounds in diabetic patients (PMID: 32633896). In this intervention technique, therapeutic concentrations of medical-grade CO2 are applied to the skin's surface in a safe, non-invasive manner. The main therapeutic mechanism is derived from the human body's natural response to locally increased CO2 concentration. Because vasodilatory capacity is impaired in diabetic foot, these mechanisms enhance local microvascular perfusion, thereby improving tissue oxygenation in patients with DFUs. Furthermore, although the researchers primarily focus on CO2 therapy as an intervention method, its efficacy is also suggested in preventing DFUs. We plan to enrole 120 patients, 80 into the study arm that will recieve CO2 therapy and 40 for a control group wothout CO2 therapy. All 120 patienrs will receive standard wound care. Aditionally, only study group will receive 20 treatments with CO2 (each workday for 4 weeks). Lower part of the body will be inserted into therapeutic wrap that is filled with 99.9% CO2 gas for 50 minutes. In both groups investigator will evaluate wound status (size, Falanga score of the wound bed) before first and after 4 weeks of treatment. Main outcome measure will be ratio of the completely heald wounds, reduction of the wound size in non healed wounds and status of the wound bed in non healed wounds after 4 weeks of treatment. Possible side effects of the CO2 therapy will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of DM Type 1 or Type 2,
* confirmed diagnosis of a non-healing DFU without clinical signs of infection,
* being able to provide informed consent for the participation, and

Exclusion Criteria:

* patients with severe comorbidities: deep vein thrombosis, chronic kidney diseases grade III and IV, chronic heart diseases NYHA (New York Heart Association) III and IV, patients with known malignant diseases, patients with progressive infection, signs of systemic infection with elevated inflammatory markers or osteomyelitis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Ratio of completely healed wounds | after 4 weeks of therapy with CO2 or standard of care
  The ratio of the completely healed wounds without exudate on 2 consecutive visits

SECONDARY OUTCOMES:
reduction of the wound size of the unhealed wounds | after 4 weeks of therapy with CO2 or standard of care
  the ratio of the reduction of the wound size in wound that are not completely helaed after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Igor Frangez, PhD, MD, DDS, Principal Investigator — UCMLjubljana
Locations (3):
- Clinical Hospital Merkur, University Clinic for Diabetes, Endocrinology, and Metabolic Diseases Vuk Vrhovac, Dugi dol 4a, 10000 Zagreb, Zagreb, Croatia, Croatia
- Slovenia (2):
  - UMCLjubljana, Ljubljana, Ljubljana
  - General hospital Novo mesto, Novo Mesto, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith AG, Ramachandran P, Tripp S, Singleton JR. Epidermal nerve innervation in impaired glucose tolerance and diabetes-associated neuropathy. Neurology. 2001 Nov 13;57(9):1701-4. doi: 10.1212/wnl.57.9.1701. PMID 11706115
- [Background] Sakai Y, Miwa M, Oe K, Ueha T, Koh A, Niikura T, Iwakura T, Lee SY, Tanaka M, Kurosaka M. A novel system for transcutaneous application of carbon dioxide causing an "artificial Bohr effect" in the human body. PLoS One. 2011;6(9):e24137. doi: 10.1371/journal.pone.0024137. Epub 2011 Sep 8. PMID 21931656
- [Background] Macura M, Ban Frangez H, Cankar K, Finzgar M, Frangez I. The effect of transcutaneous application of gaseous CO2 on diabetic chronic wound healing-A double-blind randomized clinical trial. Int Wound J. 2020 Dec;17(6):1607-1614. doi: 10.1111/iwj.13436. Epub 2020 Jul 7. PMID 32633896
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709